CLINICAL TRIAL: NCT07058857
Title: The Effect of Low-Level Tragus Stimulation on Echocardiographic Parameters in Patients With ST-Segment Elevation Myocardial Infarction - A Single-Centre Randomized Control Trial
Acronym: ELITE-STEMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Diponegoro (Other)
Responsible Party: Principal Investigator, Sodiqur Rifqi, Principal Investigator; Former of Head of Department of Cardiovascular Medicine Faculty of Medicine Universitas Diponegoro, Universitas Diponegoro
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Undip_Kardio 5
Record Dates: First submitted 2025-06-30; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: ST-segment elevation myocardial infarction; Low level tragus stimulation; Left ventricular ejection fraction; Wall motion score index
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant will not know either they include in treatment or control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low Level Tragus Stimulation Group (Experimental): Participant will undergo low level tragus stimulation using Parasym Device
  Interventions: Device: Parasym Neuromodulation Device (Treatment Group); Device: Parasym Neuromodulation Device (Sham Group)
- Sham Control Group (Sham Comparator): Participant will have Parasym Device implanted in their tragus without any active stimulation from the device
  Interventions: Device: Parasym Neuromodulation Device (Treatment Group); Device: Parasym Neuromodulation Device (Sham Group)

INTERVENTIONS:
Device: Parasym Neuromodulation Device (Treatment Group) — Participant will undergo stimulation in their left tragus for 60 minutes by using Parasym device
Device: Parasym Neuromodulation Device (Sham Group) — Participant will undergo implantation of Parasym device lead in their left tragus but without any stimulation for 60 minutes

SUMMARY:
The goal of this clinical trial is to learn the effect of low level tragus stimulation (LLTS) on echocardiographic parameter in patient with ST-segment Elevation Myocardial Infarction (STEMI) who undergo primart percutaneous coronary intervention (PPCI). It will also learn about the safety of LLTS in such setting. The main questions, it aims to answer are compared with sham control:

Does LLTS could alter left ventricular ejection fraction in patients with STEMI? Does LLTS could alter wall motion score index in patients with STEMI? Does LLTS could alter diastolic dysfunction in patients with STEMI?

Researchers will compare LLTS to sham LLTS control to see if LLTS have benefit in participants with STEMI participants will divided into two group i.e. treatment group vs control (sham/placebo) group..

Both groups undergo transthoracal echocardiographi examination before and after PPCI..

ELIGIBILITY:
Inclusion Criteria:

* Onset STEMI less than 12 hours
* Participant agreed to be included in this study
* Killip class I - II on presentation
* SBP >90 mmHg and/or MAP >65 mmHg
* Sinus rhtyhm

Exclusion Criteria:

* History of myocardial infarction, stroke, heart failure with reduce ejection fraction, chronic total occlussion on prior coronary angiography, chronic kidney disease (eGFR < 30) or on hemodyalisis, malignancy, hematology disease, autoimmune, or other chronic diseases
* On permanent pacemaker
* Acute infection
* Pregnant woman

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Left Ventricular Ejection Fraction | Before PPCI, 1 day after PPCI, and 30 days after PPCI
  Left Ventricular Ejection Fraction measured by transthoracic echocardiography

SECONDARY OUTCOMES:
Wall Motion Score Index | Before PPCI, 1 day after PPCI, and 30 days after PPCI
  Wall Motion Score Index measured by transthoracic echocardiography
Diastolic Function | Before PPCI, 1 day after PPCI, and 30 days after PPCI
  Diastolic Function measured by transthoracic echocardiography

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Kariadi Central General Hospital, Semarang, Central of Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yu L, Huang B, Po SS, Tan T, Wang M, Zhou L, Meng G, Yuan S, Zhou X, Li X, Wang Z, Wang S, Jiang H. Low-Level Tragus Stimulation for the Treatment of Ischemia and Reperfusion Injury in Patients With ST-Segment Elevation Myocardial Infarction: A Proof-of-Concept Study. JACC Cardiovasc Interv. 2017 Aug 14;10(15):1511-1520. doi: 10.1016/j.jcin.2017.04.036. PMID 28797427
- [Background] Redgrave J, Day D, Leung H, Laud PJ, Ali A, Lindert R, Majid A. Safety and tolerability of Transcutaneous Vagus Nerve stimulation in humans; a systematic review. Brain Stimul. 2018 Nov-Dec;11(6):1225-1238. doi: 10.1016/j.brs.2018.08.010. Epub 2018 Aug 23. PMID 30217648